CLINICAL TRIAL: NCT06576466
Title: Effect of Supplementation With Creatine on the Early Recovery of Ischemic Stroke: A Randomized Clinical Trial
Brief Title: Effect of Supplementation With Creatine on the Recovery of Ischemic Stroke
Acronym: SUCRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Collaborators: Comunidad Autónoma de las Islas Baleares (Dirección General de Investigación en Salud, Formación y Acreditación) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROSALUT2023-27
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-07

CONDITIONS: Stroke, Ischemic
Keywords: stroke; creatine; sarcopenia
MeSH Terms: conditions — Ischemic Stroke; Stroke; Sarcopenia | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A professional from the pharmacy service, who will not be involved in data collection or participant care, will handle the blinding.
  The care staff responsible for patient care will be unaware of each participant's assignment group.
  Blinding may be broken if a serious adverse effect related to the supplementation is suspected in one of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Creatine monohydrate (Experimental): Creatine monohydrate. Guinama brand with CE marking. Code 89823.
  Interventions: Dietary Supplement: Creatine monohydrate
- Dextromaltose (Placebo Comparator): Dextrinomaltose. Guinama brand with CE marking. Code 91146.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — Creatine monohydrate. Guinama brand with CE marking. Code 89823.
  Arms: Creatine monohydrate
Other: Placebo — Dextrinomaltose. Guinama brand with CE marking. Code 91146.
  Arms: Dextromaltose

SUMMARY:
Stroke is a leading cause of disability and the second leading cause of death worldwide. Most strokes are ischemic, caused by acute arterial occlusion. Post-stroke treatment focuses on secondary prevention and rehabilitation, but few treatments address functional recovery. Creatine, a supplement known for improving physical performance, may aid in the recovery of stroke patients, reducing sarcopenia and improving strength among other effects. This pilot study will investigate the effectiveness of creatine supplementation in enhancing physical and functional recovery in ischemic stroke patients. The study will involve a randomized, double-blind clinical trial comparing creatine monohydrate to a placebo.

DETAILED DESCRIPTION:
Stroke is one of the most impactful health conditions worldwide, currently being the leading cause of disability and the second leading cause of death globally. Approximately 85-90% of strokes are ischemic, primarily caused by acute arterial occlusion, leading to an area of cerebral, spinal, or retinal infarction. The size of the lesion depends on the affected blood vessel and the duration of the occlusion, as well as cerebral autoregulation, blood pressure, blood sugar levels, and many other factors. After the acute phase, treatment is based on secondary prevention and rehabilitation, with few treatments currently available that focus on functional recovery once the infarction has occurred. Stroke survivors experience a loss of functionality, a decline in physical capacity associated with a decrease in muscle mass, sarcopenia, cognitive impairment, and an increase in anxiety and depressive symptoms.

Creatine is a widely studied nutritional supplement, mainly in athletes, where it has been shown to improve training adaptation and physical performance. Its effects on energy metabolism, as an anti-inflammatory, and on calcium homeostasis have been described. There are also studies indicating possible musculoskeletal benefits in the elderly population. Given its role in improving physical performance and muscle mass, considering the significant impact of these conditions on patients who have suffered an ischemic stroke, and considering its antioxidant and anti-inflammatory effects, we propose a pilot study to determine the effectiveness of creatine supplementation in stroke patients. This supplementation could potentially lead to greater physical and functional recovery following an ischemic stroke.

A randomized, double-blind clinical trial will be conducted. The trial will include a group supplemented with creatine monohydrate at a dose of 0.3 g/kg/day for 7 days, followed by 0.1 g/kg/day for 12 weeks, alongside standard clinical practice; and a control group supplemented with a placebo (corn starch maltodextrin), following the same protocol and doses.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Recent diagnosis of ischemic stroke (from 24 hours to 5 days) .
* Neurological deficit due to the stroke that affects mobility (paresis and/or ataxia) and requires motor rehabilitation.
* Ability to understand and sign the informed consent form, or failing that, have sufficient support to carry out the correct follow-up of the study.

Exclusion Criteria:

* Moderate-severe disability prior to stroke, defined by an mRS>2.
* Unstable or severe clinical situation that prevents active rehabilitation.
* Neurological deficit due to stroke that prevents walking without help from another person. The use of support with a cane, crutch or walker is permitted.
* Moderate or severe dysphagia that makes therapeutic adherence difficult.
* Use of creatine supplements in the last 3 months, or use of anabolic products in the last 3 months.
* Severe kidney disease (GFR <30ml/min/1.73 m2).
* Musculoskeletal pathology that prevents assessment of muscle strength. For example: fractures, severe osteoarthritis, ligament tears or tendinopathies.
* History of allergic reactions to creatine.
* Pregnancy or breastfeeding.
* Simultaneous participation in another clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Physical performance | 3 months, 6 months
  To analyze the improvement in physical performance, at 3 months (at the end of the intervention) and at 6 months, measured by the 6-Minute Walking Test (6MW).

SECONDARY OUTCOMES:
Physical performance using Test "timed up and go" (TUG). | 3 months, 6 months
  Test "timed up and go" (TUG).
Maximum muscle strength | 3 months, 6 months
  Maximum muscle strength, measured by manual dynamometer (Kilograms). Grip strength, biceps, triceps, deltoids, psoas, quadriceps and hamstrings will be assessed.
Arm and leg muscle strength | 3 months, 6 months
  Measured by the score on items 5 and 6 of the National institute of Health Stroke Scale (NIHSS) where the score range is from 0 to 4. A higher score corresponds to a worse performance.
Balance and stability | 3 months, 6 months
  Balance and stability measured using the Postural Assessment Scale for Stroke Patients (PASS). The scale includes 12 items, which are divided into two categories: maintaining a posture (static balance) and changing a posture (dynamic balance). Higher scores indicate better postural control and balance.
Functional impact | 3 months, 6 months
  Functional impact measured by the Modified Rankin Scale (mRS). The mRS is a commonly used scale to measure the degree of disability or dependence in daily activities of people who have suffered a stroke. The mRS is scored on a scale from 0 to 6, with higher scores indicating greater disability
Performance in basic activities of daily living | 3 and 6 months
  Barthel Scale. The Barthel Index is a scale used to measure a person's performance in basic activities of daily living (ADLs) and assess functional independence
Cognitive assessment | 3 months
  Cognitive assessment using the Montreal cognitive assessment (MoCA) test. The MoCA is a tool used to assess cognitive impairment in various domains, including memory, attention, language, and executive function. A higher score means a better outcome.
Quality of life measured by EuroQol 5D | 3 months, 6 months
  Quality of life assessment using the "EuroQol 5D". EuroQoL 5D is a standardized tool used to assess health-related quality of life. A higher score corresponds to worse quality of life.
Anxiety and depression symptoms | 3 months
  Assessment of anxiety and depression symptoms using the HADS (Hospital Anxiety and Depression Scale). Both the Anxiety subscale and the Depression subscale range from 0 to 21. Higher scores on either subscale indicate worse outcomes (more severe anxiety or depression).
Appendicular skeletal muscle mass | 3 months
  Measurement of appendicular (arms and legs) skeletal muscle mass change from baseline, using DXA (dual-energy X-ray absorptiometry) measured in kilograms. A higher skeletal muscle mass means a better outcome.
Total skeletal muscle mass | 3 months
  Measurement of total skeletal muscle mass change from baseline, using DXA (dual-energy X-ray absorptiometry) measured in kilograms. A higher skeletal muscle mass means a better outcome.
Appendicular body fat | 3 months
  Measurement of appendicular (arms and legs) and total body fat change from baseline, using DXA (dual-energy X-ray absorptiometry) measured in kilograms. A lower fat mass means a better outcome.
Total body fat | 3 months
  Measurement of total body fat change from baseline, using DXA (dual-energy X-ray absorptiometry) measured in kilograms. A lower fat mass means a better outcome.
Nutritional status | 3 months, 6 months
  Measurement of nutritional status change by phase angle using a bioelectrical impedance analysis. A higher phase angle means a better outcome. Outcome units are degrees.
Number of falls. | 3 months, 6 months
  Number of falls since last visit.
Geriatric Nutritional Risk Index (GNRI) score | 3 months, 6 months
  Geriatric Nutritional Risk Index (GNRI) score. The following formula is used: [1.489 × serum albumin (g/L)] + (41.7 × weight (kg)/ideal weight (kg)).
Ventricular strain change | 3 months
  Effect of creatine on cardiac damage secondary to stroke measured using ventricular strain measurement (percentage). A lower strain corresponds to a worse outcome.
Ejection fraction change | 3 months
  Effect of creatine on cardiac damage secondary to stroke measured using ejection fraction (EF) measurement (percentage). A lower EF corresponds to a worse outcome.
Adverse events | From enrollment to the end of treatment at 6 months
  To assess the occurrence of any adverse events in any of the intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Delgado Mederos, PhD, Principal Investigator — Fundació d'investigació Sanitària de les Illes Balears
Locations (1):
- IdISBa, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in Creatine supplementation and stroke. Data will be shared subject to acceptance by the research team. Data or samples shared will be coded.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 24 months.
Access Criteria: Access to trial IPD can be requested by qualified researchers. Data will be shared subject to acceptance by the research team.

REFERENCES:
- [Background] Bender A, Samtleben W, Elstner M, Klopstock T. Long-term creatine supplementation is safe in aged patients with Parkinson disease. Nutr Res. 2008 Mar;28(3):172-8. doi: 10.1016/j.nutres.2008.01.001. PMID 19083405
- [Background] Gualano B, de Salles Painelli V, Roschel H, Lugaresi R, Dorea E, Artioli GG, Lima FR, da Silva ME, Cunha MR, Seguro AC, Shimizu MH, Otaduy MC, Sapienza MT, da Costa Leite C, Bonfa E, Lancha Junior AH. Creatine supplementation does not impair kidney function in type 2 diabetic patients: a randomized, double-blind, placebo-controlled, clinical trial. Eur J Appl Physiol. 2011 May;111(5):749-56. doi: 10.1007/s00421-010-1676-3. Epub 2010 Oct 26. PMID 20976468
- [Background] Pan JW, Takahashi K. Cerebral energetic effects of creatine supplementation in humans. Am J Physiol Regul Integr Comp Physiol. 2007 Apr;292(4):R1745-50. doi: 10.1152/ajpregu.00717.2006. Epub 2006 Dec 21. PMID 17185404
- [Background] McMorris T, Mielcarz G, Harris RC, Swain JP, Howard A. Creatine supplementation and cognitive performance in elderly individuals. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2007 Sep;14(5):517-28. doi: 10.1080/13825580600788100. PMID 17828627
- [Background] Turner CE, Byblow WD, Gant N. Creatine supplementation enhances corticomotor excitability and cognitive performance during oxygen deprivation. J Neurosci. 2015 Jan 28;35(4):1773-80. doi: 10.1523/JNEUROSCI.3113-14.2015. PMID 25632150
- [Background] Butchart S, Candow DG, Forbes SC, Mang CS, Gordon JJ, Ko J, Deprez D, Chilibeck PD, Ditor DS. Effects of Creatine Supplementation and Progressive Resistance Training in Stroke Survivors. Int J Exerc Sci. 2022 Aug 1;15(2):1117-1132. doi: 10.70252/EKHJ1489. eCollection 2022. PMID 35992184
- [Background] Forbes SC, Cordingley DM, Cornish SM, Gualano B, Roschel H, Ostojic SM, Rawson ES, Roy BD, Prokopidis K, Giannos P, Candow DG. Effects of Creatine Supplementation on Brain Function and Health. Nutrients. 2022 Feb 22;14(5):921. doi: 10.3390/nu14050921. PMID 35267907
- [Background] Solis MY, Artioli GG, Otaduy MCG, Leite CDC, Arruda W, Veiga RR, Gualano B. Effect of age, diet, and tissue type on PCr response to creatine supplementation. J Appl Physiol (1985). 2017 Aug 1;123(2):407-414. doi: 10.1152/japplphysiol.00248.2017. Epub 2017 Jun 1. PMID 28572496
- [Background] Chrusch MJ, Chilibeck PD, Chad KE, Davison KS, Burke DG. Creatine supplementation combined with resistance training in older men. Med Sci Sports Exerc. 2001 Dec;33(12):2111-7. doi: 10.1097/00005768-200112000-00021. PMID 11740307
- [Background] Scherbakov N, von Haehling S, Anker SD, Dirnagl U, Doehner W. Stroke induced Sarcopenia: muscle wasting and disability after stroke. Int J Cardiol. 2013 Dec 10;170(2):89-94. doi: 10.1016/j.ijcard.2013.10.031. Epub 2013 Oct 14. PMID 24231058
- [Background] Coleman ER, Moudgal R, Lang K, Hyacinth HI, Awosika OO, Kissela BM, Feng W. Early Rehabilitation After Stroke: a Narrative Review. Curr Atheroscler Rep. 2017 Nov 7;19(12):59. doi: 10.1007/s11883-017-0686-6. PMID 29116473
- [Background] Balestrino M. Role of Creatine in the Heart: Health and Disease. Nutrients. 2021 Apr 7;13(4):1215. doi: 10.3390/nu13041215. PMID 33917009
- [Background] Schroder H, Fito M, Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Lamuela-Raventos R, Ros E, Salaverria I, Fiol M, Lapetra J, Vinyoles E, Gomez-Gracia E, Lahoz C, Serra-Majem L, Pinto X, Ruiz-Gutierrez V, Covas MI. A short screener is valid for assessing Mediterranean diet adherence among older Spanish men and women. J Nutr. 2011 Jun;141(6):1140-5. doi: 10.3945/jn.110.135566. Epub 2011 Apr 20. PMID 21508208
- [Background] Scheitz JF, Sposato LA, Schulz-Menger J, Nolte CH, Backs J, Endres M. Stroke-Heart Syndrome: Recent Advances and Challenges. J Am Heart Assoc. 2022 Sep 6;11(17):e026528. doi: 10.1161/JAHA.122.026528. Epub 2022 Sep 3. PMID 36056731
- See also: Stroke among top 10 causes of death according to the Word Health Organization (WHO). — http://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death